CLINICAL TRIAL: NCT03174093
Title: A Mobile Health Application to Improve Anticoagulation Care in Atrial Fibrillation: Randomized Controlled Trial
Brief Title: Mhealth Application for anTicoagulation Care in Atrial Fibrillation
Acronym: MATCh AFib
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Instituto de Cardiologia do Rio Grande do Sul (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 5043/14
Record Dates: First submitted 2017-01-18; First posted 2017-06-02 (Actual); Last update posted 2017-06-02 (Actual); Status verified 2017-06

CONDITIONS: Atrial Fibrillation; Anticoagulants; Circulating, Hemorrhagic Disorder
Keywords: Mobile Health
MeSH Terms: conditions — Atrial Fibrillation; Hemorrhagic Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MATCh AFib (Experimental): Participants assigned to the intervention group will have the support of the MATCh AFib application during the consultations with their physician and receive individual text messaging targeting knowledge about atrial fibrillation, medication adherence and monitoring during months 1-3.
  Interventions: Behavioral: MATCh AFib application
- Standard Care (No Intervention): Participants assigned to the control group will complete measures at each time point and maintain care as usual (i.e., medical treatment, INR monitoring and consultations with their physician without mHealth support)

INTERVENTIONS:
Behavioral: MATCh AFib application — The application comprehends five steps: (1) An educational video about how AF can cause stroke; (2) A calculator of risk scores (CHA2DS2-VASc, HAS-BLED and SAMe-TT2R2); (3) A screen with pictograms to allow better understanding of the scores by patients and to demonstrate how much each anticoagulant can decrease stroke risk or increase bleeding risk; (4) A summary about types of medications available, and (5) An output formulary in which the physician can register patient's contact to continue receiving information about atrial fibrillation and anticoagulation through SMS. Physicians can save patient's history of INR tests and previous doses of anticoagulation prescribed and also use a calculator to adjust the dose.
  Arms: MATCh AFib

SUMMARY:
This study will assess the benefits of using a mobile health application designed for shared decision aid in anticoagulation therapy in patients with Atrial Fibrillation (AF). The aim is to improve their treatment adherence and time in therapeutic International Normalized Ratio (INR) range. The results of this study have the potential to lead to a sustainable and resource-efficient strategy for better prevent thromboembolic events in patients with atrial fibrillation.

DETAILED DESCRIPTION:
Atrial Fibrillation is a common disease, with important burden on morbidity and mortality and a challenging management. Its incidence and healthcare costs have increased over the decades. One of the most important features of this arrhythmia is its stroke risk, which can be reduced with the use of anticoagulants. Deciding about anticoagulation therapy is complicated due to frequent competing comorbidities and potential harms of the therapy itself. To achieve better outcomes in preventing stroke, it is paramount that decisions about atrial fibrillation treatment be shared between providers and patients.

Mobile health is empowering individuals to assume a more active role in monitoring and managing their chronic conditions and therapeutic regimens. Also, health professionals are being provided with fast and point-of-care information, which can facilitate decision-making.

Therefore, this study will investigate the effects of an mHealth application idealized to aid shared decision and improve anticoagulation care in atrial fibrillation.

Adults with atrial fibrillation will be recruited from anticoagulation outpatient clinics and Basic Health Units and randomized to either (1) an intervention group in which the mHealth application will be used during the consultations or (2) a control group receiving the usual care with anticoagulation.

It is hypothesized that the intervention group will achieve better anticoagulation outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Adults >=18 years
* Diagnostic of atrial fibrillation
* Indication of oral anticoagulation by their physician, based on risk scores
* Ability to speak, hear and understand Portuguese
* Able to receive and read text messages through a cell phone

Exclusion Criteria:

Physical impairments that prevent completion of the intervention, cognitive impairments that jeopardize informed consent and/or intervention comprehension and not fluent in Portuguese.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2017-06 (Estimated); Primary Completion 2018-06 (Estimated); Study Completion 2018-11 (Estimated)

PRIMARY OUTCOMES:
Oral anticoagulant adherence | 6 months
  For patients on Non-vitamin K antagonists oral anticoagulants, a change from baseline in oral anticoagulant adherence at 6 months to achieve a percentage of days covered (PDC) from 50% to 80%.
Percent time in therapeutic INR (TTR) | 6 months
  For patients on Vitamin-K antagonists, a change from baseline in TTR at 6 months from 50% to 60%.
  TTR: percent time in therapeutic INR range calculated by Rosendaal method. An INR value of >2.0 was defined as subtherapeutic, and an INR value <3.0 was defined as supratherapeutic.

SECONDARY OUTCOMES:
Decisional Conflict Scale | After decision about anticoagulant usually 30 minutes after consultation and on study completion (6 months)
  Personal perception of decisional conflict measured by the Decisional Conflict Scale (DCS) of O'Connor

IPD SHARING:
Plan to Share IPD: No